CLINICAL TRIAL: NCT07152938
Title: The Effect of Using Augmented Virtual Reality on Pain, Stress, Anxiety, and Self-Efficacy Among Adult Cancer Patients Undergoing Chemotherapy in the West Bank
Brief Title: Augmented Virtual Reality for Reducing Pain, Stress, Anxiety and Improve Self Efficacy in Adult Cancer Patients Undergoing Chemotherapy in The West Bank
Acronym: AVR-CHEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Farid Salih Abu lie, academic lecturer, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAUP-AVR-ONCO-2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cancer and Chemotherapy Related Anemia; Cancer (Colon Cancer, Breast Cancer, Lymphoma, Chronic Lymphoma Leukemia, Multiple Myeloma)
Keywords: Augmented Virtual Reality; Pain Management; Stress; Anxiety; Self-Efficacy; Chemotherapy; Palestine
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lymphoma; Multiple Myeloma; Agnosia; Anxiety Disorders | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: participants randomly assigned to either the intervention group(augmented virtual reality sessions)or the other control group( standard care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Chemotherapy Care) (No Intervention): the control group participated in routine sessions without AVR. Patients were admitted to the daycare unit, where a cannula was applied. The nurse then followed the doctor's order for the type of medication that would be given to the patient. Subsequently, the patients filled out the questionnaire at the posttest.
- AVR Group (Experimental): Patients receive standard chemotherapy care plus Augmented Virtual Reality (AVR) distraction sessions during chemotherapy infusion.
  Interventions: Behavioral: AVR Group (Chemotherapy + AVR)

INTERVENTIONS:
Behavioral: AVR Group (Chemotherapy + AVR) — the intervention group received AVR before they started treatment and during the session. The researcher administered the posttest questionnaire The questionnaire assessed immediately after finishing AVR. Participants informed not to discuss AVR with each other's, as the researcher explained to the participants the purpose of the study and their participation will not affect their care or treatment
  Arms: AVR Group

SUMMARY:
The main purpose of this study is to examine the effect of using AVR on pain, stress, anxiety, and SE among adult cancer patients undergoing chemotherapy in the West Bank hospitals in Palestine. The main questions it aims to answer are:

1. What is the effect of AVR therapy on pain levels score compared with routine care during chemotherapy session among cancer patients?
2. What is the effect of AVR therapy on the stress levels compared with routine care during chemotherapy session among cancer patients?
3. What is the effect of AVR therapy on the anxiety compared with routine care during chemotherapy session among cancer patients?
4. What is the effect of AVR therapy on the general SE compared with routine care during chemotherapy session among cancer patients?

The participants divided into two groups, the intervention group, which receives AVR, and the control group, which receives standard treatment. The study used a pretest and posttest design to assess the effect of AVR on the study variables (pain, stress, anxiety and self-efficacy).

DETAILED DESCRIPTION:
This study was designed as a randomized control trial (RCT), including both pretest and posttest assessments.

Participants were randomly assigned to either the intervention group, which received AR, or the control group, which received standard treatment. Random assignment was conducted using a computer-generated list of patients scheduled for chemotherapy, with patients alternately assigned to the intervention and control group (e.g., patient number 1 to the intervention group, number 2 to the control group). This process was managed by a nurse who was blinded to the study protocol. Due to the nature of the study, the researchers were not blinded.

The study was conducted in three large hospitals in northern Palestine that specialized in oncology care, particularly within their chemotherapy units.

The sample consisted of cancer patients undergoing chemotherapy in the aforementioned hospitals. Pretests, interventions, and posts were conducted .Inclusion criteria were cancer patients (over 18 years old) who required chemotherapy and could provide informed consent in Arabic. Exclusion criteria included a history of VR motion sickness, physical or cognitive limitations preventing VR headset use, visual, auditory, or vestibular impairments, uncontrolled severe medical conditions (e.g., vomiting, nausea, respiratory depression), pediatric patients, cognitive impairments, and any mental or psychological disorders.

Questionnaires were used to gather the data. It consists of three sections:

Sociodemographic data: composed of age gender, resident area, marital status, type of cancer, number of chemotherapy sessions, and medical data

the variables assessed used the below tool

1. Numeric Pain Rating Scale (NPRS):

   This scale was developed for assessing the pain scale.
2. Perceived Stress Scale (PSS-10) The Perceived Stress Scale (PSS-10)
3. Generalized Anxiety disorder (GAD-7) The GAD-7 A brief measure for assessing generalized anxiety disorder: the GAD-7.
4. General Self-Efficacy Scale (GSE) The scale is designed to assess a person's optimistic self-beliefs used to cope with life's demands

Data Collection Process Data were collected from June to September 2023. Ethical approval was obtained from the Arab American University and the Palestinian Ministry of Health. The data collection process began with a meeting with the head of the chemotherapy unit to compile a list of eligible patients. Randomization ensured equal chance of participants for all eligible patients

The study was conducted in two phases to prevent contamination between groups:

Phase one (Control Group): Patients received routine chemotherapy sessions without VR. Before and after the sessions, they completed the pre and post-test questionnaires.

Phase two (Intervention Group): patients received VR during their chemotherapy sessions. Pre and post-test questionnaires were administered before and after the VR sessions.

Both groups completed the questionnaires during their regular visits to the chemotherapy units. The post-intervention assessment measured levels of stress and anxiety using the same questionnaires as the pretest.

Once participants prepared for chemotherapy infusion, investigator provided them with the VR headset with a brief overview of how the hardware worked. This includes details on how to navigate the interface, and which apps were available for use during the intervention. Participants completed a brief survey through a self-administered questionnaire to assess their levels of stress and anxiety. The participants chose to experience which video they would like to watch mountains, rivers, sea, and mountain falls.

Participants were provided with a Meta Quest 2 headset (KW49CM), equipped with high-resolution displays and paired with the Meta-Quest iOS app (version 192.0). Patients were given a brief overview of how to use the hardware and could choose from soothing virtual environments such as mountains, rivers, and waterfalls.

A pilot study was conducted on 15 patients meeting the study criteria. The pilot aimed to test the feasibility and reliability of the study design.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-60 years undergoing chemotherapy for breast or colon cancer.
2. Stage I or II cancer, as defined by the study protocol.
3. Manageable levels of pain, anxiety, and stress, appropriate for participation in the intervention.

   -

Exclusion Criteria:

1. Age over 60 years.
2. Cancer types other than breast or colon cancer.
3. Severe pain, anxiety, or stress that could interfere with participation or require intensive care beyond the study scope.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity during chemotherapy | Immediately before chemotherapy and immediately after the session (June 2023 - September 2023).
  Pain intensity will be measured using the Numeric Pain Rating Scale (NPRS). The NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater pain intensity. The outcome will be the change in NPRS score from immediately before to immediately after the chemotherapy session, comparing the AVR intervention group with the control group.

SECONDARY OUTCOMES:
Change in self-efficacy during chemotherapy | Immediately before chemotherapy and immediately after the session (June 2023 - September 2023).
  Self-efficacy will be measured using the General Self-Efficacy Scale (GSE). The GSE consists of 10 items, each scored from 1 (not at all true) to 4 (exactly true), with total scores ranging from 10 to 40. Higher scores indicate greater self-efficacy. The outcome will be the change in GSE score from immediately before to immediately after the chemotherapy session, comparing the AVR intervention group with the control group.
Change in perceived stress during chemotherapy | Immediately before chemotherapy and immediately after the session (June 2023 - September 2023).
  Stress will be measured using the Perceived Stress Scale (PSS-10). The PSS-10 consists of 10 items, each scored from 0 (never) to 4 (very often), with total scores ranging from 0 to 40. Higher scores indicate greater perceived stress. The outcome will be the change in PSS-10 score from immediately before to immediately after the chemotherapy session, comparing the AVR intervention group with the control group.
Change in anxiety symptoms during chemotherapy | Immediately before chemotherapy and immediately after the session (June 2023 - September 2023).
  Anxiety will be measured using the Generalized Anxiety Disorder Scale (GAD-7). The GAD-7 consists of 7 items, each scored from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptoms. The outcome will be the change in GAD-7 score from immediately before to immediately after the chemotherapy session, comparing the AVR intervention group with the control group.

CONTACTS AND LOCATIONS:
Locations (3):
- Palestinian Territories (3):
  - Jenin governmental hospital, Jenin
  - AL-Watni governmental hospital, Nablus
  - Thabet Thabet governmental hospital, Tulkarm

IPD SHARING:
Plan to Share IPD: No
Individual participant data did not shared due to patient privacy concerns and the absence of a secure data repository. Only aggregated and anonymized study results made available in publications and presentations